CLINICAL TRIAL: NCT01418209
Title: MsFLASH-03: Comparative Efficacy of Low-Dose Estradiol and the SNRI Venlafaxine XR for Treatment of Menopausal Symptoms
Brief Title: MsFLASH-03: Comparative Efficacy of Low-Dose Estradiol and Venlafaxine XR for Treatment of Menopausal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); Office of Research on Women's Health (ORWH) (NIH)
Responsible Party: Principal Investigator, Katherine Guthrie, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MsFLASH-03; 1U01AG032700-01 (NIH); 1U01AG032699-01 (NIH)
Record Dates: First submitted 2011-08-15; First posted 2011-08-17 (Estimated); Results first posted 2014-08-20 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Hot Flashes; Menopause; Vasomotor Disturbance
Keywords: Menopause; Vasomotor; Symptoms; Estradiol; Venlafaxine
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low-dose 17-ß-estradiol with progesterone taper (Active Comparator)
  Interventions: Drug: Low-dose 17-ß-estradiol with progesterone taper
- Venlafaxine XR (Active Comparator)
  Interventions: Drug: Venlafaxine XR
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low-dose 17-ß-estradiol with progesterone taper — Low-dose 17-ß-estradiol oral (by mouth), 0.5 mg once per day for 8 (eight) weeks. 17-ß-estradiol is approved by the US Food and Drug Administration (FDA) and is indicated for the treatment of menopausal symptoms. ß is the Greek symbol for beta; the symbol and the word are used interchangeably. The 8 week estradiol treatment is followed by 14 days (2 weeks) of progesterone taper (as medroxy-progesterone 10 mg/day).
  Other Names: The brand name of estradiol being used in this study is Estrace®.
  Arms: Low-dose 17-ß-estradiol with progesterone taper
Drug: Venlafaxine XR — Venlafaxine oral (by mouth) 37.5 mg once per day for 1 (one) week, then 75 mg once per day for 7 (seven) weeks. Venlafaxine XR should not be taken while also taking monoamine oxidase inhibitors (MAOIs). Venlafaxine XR is approved by the US Food and Drug Administration (FDA) for treatment of depression, generalized anxiety disorder, social anxiety disorder, and panic disorder, and is available by prescription. Venlafaxine XR is not FDA-approved for the treatment of hot flashes, although prior studies have indicated that it is useful for treating hot flashes and vasomotor symptoms. After the 8-week venlafaxine XR study treatment period, women will receive a tapering dose of venlafaxine XR 37.5 mg once per day for 14 days (2 weeks).
  Other Names: The brand name of venlafaxine XR that is being used in this study is Effexor XR®
  Arms: Venlafaxine XR
Drug: Placebo — The placebo is an inactive pill that looks like the active medication.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine the efficacy of both low-dose oral (by mouth) 17-ß-estradiol and the non-hormonal drug venlafaxine XR compared to placebo in reducing hot flashes. Included in this objective is the intention to compare venlafaxine XR to estradiol therapy, to provide evidence of the relative efficacy of venlafaxine to what is currently considered the most established but also a controversial therapy. 17-ß-estradiol is a type of estrogen. Venlafaxine XR is the extended release (XR) version of venlafaxine. Venlafaxine XR is an serotonin-norepinephrine reuptake inhibitor (SNRI). A placebo is a substance containing no medication.

DETAILED DESCRIPTION:
The MsFLASH-03 study (Menopausal Strategies: Finding Lasting Answers for Symptoms and Health - 03), Comparative Efficacy of Low-Dose Estradiol and the SNRI Venlafaxine XR for Treatment of Menopausal Symptoms, is a randomized, double-blind, placebo-controlled, three arm clinical trial. The design includes: 3 weeks of daily recording of hot flashes prior to drug treatment; 8 weeks of double-blind treatment with oral estradiol, venlafaxine, or placebo; followed by 14 days of drug taper for those on venlafaxine and 14 days of progesterone treatment for those on estradiol; followed by 2 weeks with no treatment for all groups; and a telephone follow-up post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 40-62 years
* Postmenopausal or perimenopausal
* Having bothersome hot flashes
* In general good health
* Signed informed consent

Exclusion Criteria:

* Recent use of systemic hormone therapy or hormonal contraceptives
* Recent use of any prescribed, over-the-counter or herbal therapies that are taken specifically for hot flashes
* Recent use of selective estrogen receptor modulators (SERMS) or aromatase inhibitors
* Recent use of psychotropic medications, including SSRIs (selective serotonin reuptake inhibitors), serotonin-norepinephrine reuptake inhibitors (SNRIs), MAOIs (monoamine oxidase inhibitors), and other antidepressants and anxiolytics.
* Known hypersensitivity or contraindications (reasons not to take) to venlafaxine, estrogen, or progestins
* Not using a medically approved method of birth control, if sexually active and not 12 or more months since last menstrual period
* Recent drug or alcohol abuse
* Lifetime diagnosis of psychosis or bipolar disorder
* Suicide attempt in the past 3 years or any current suicidal ideation
* Current major depression (assessed during screening)
* Pregnancy, intending pregnancy, or breast feeding
* History of:

  * Pre-breast cancer or high-risk breast cancer condition
  * Abnormal bleeding suggestive of endometrial pre-cancer or endometrial hyperplasia
  * Asthma, diabetes mellitus, epilepsy, and migraine disorders that are not stable or under medical management
* Abnormal screening blood tests
* Current participation in another drug trial or intervention study
* Inability or unwillingness to complete the study procedures

Ages: 40 Years to 62 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 339 (Actual)
Dates: Start 2011-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Z LaCroix, PhD, Principal Investigator — Fred Hutchinson Cancer Center; Garnet Anderson, PhD, Principal Investigator — Fred Hutchinson Cancer Center; Katherine Guthrie, PhD, Principal Investigator — Fred Hutchinson Cancer Center; Lee S Cohen, MD, Principal Investigator — Massachusetts General Hospital/Harvard Medical School (HU); Hadine Joffe, MD, MSc, Principal Investigator — Massachusetts General Hospital/Harvard Medical School (HU); Katherine M Newton, PhD, Principal Investigator — Group Health Research Institute (GHRI); Susan D Reed, MD, Principal Investigator — University of Washington/Group Health Research Institute (GHRI); Janet Carpenter, PhD, RN, FAAN, Study Director — Indiana University School of Medicine; Ellen W Freeman, PhD, Principal Investigator — University of Pennsylvania School of Medicine (UP)
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Harvard Medical School (HU), Boston, Massachusetts
  - Brigham and Women's Hospital, Chestnut Hill, Massachusetts
  - University of Pennsylvania, UP, Philadelphia, Pennsylvania
  - Group Health Research Institute (GHRI), Seattle, Washington

REFERENCES:
- [Derived] Ensrud KE, Larson JC, Guthrie KA, Crandall CJ, LaCroix AZ, Reed SD, Bhasin S, Mitchell CM, Joffe H. Changes in serum endogenous estrogen concentrations are mediators of the effect of low-dose oral estradiol on vasomotor symptoms. Menopause. 2022 Sep 1;29(9):1014-1020. doi: 10.1097/GME.0000000000002026. Epub 2022 Aug 16. PMID 35969887
- [Derived] Hudson PL, Ling W, Wu MC, Hayward MR, Mitchell AJ, Larson J, Guthrie KA, Reed SD, Kwon DS, Mitchell CM. Comparison of the Vaginal Microbiota in Postmenopausal Black and White Women. J Infect Dis. 2021 Dec 1;224(11):1945-1949. doi: 10.1093/infdis/jiaa780. PMID 33367735
- [Derived] Diem SJ, LaCroix AZ, Reed SD, Larson JC, Newton KM, Ensrud KE, Woods NF, Guthrie KA. Effects of pharmacologic and nonpharmacologic interventions on menopause-related quality of life: a pooled analysis of individual participant data from four MsFLASH trials. Menopause. 2020 Oct;27(10):1126-1136. doi: 10.1097/GME.0000000000001597. PMID 32701665
- [Derived] Mitchell CM, Srinivasan S, Plantinga A, Wu MC, Reed SD, Guthrie KA, LaCroix AZ, Fiedler T, Munch M, Liu C, Hoffman NG, Blair IA, Newton K, Freeman EW, Joffe H, Cohen L, Fredricks DN. Associations between improvement in genitourinary symptoms of menopause and changes in the vaginal ecosystem. Menopause. 2018 May;25(5):500-507. doi: 10.1097/GME.0000000000001037. PMID 29206774
- [Derived] Guthrie KA, Larson JC, Ensrud KE, Anderson GL, Carpenter JS, Freeman EW, Joffe H, LaCroix AZ, Manson JE, Morin CM, Newton KM, Otte J, Reed SD, McCurry SM. Effects of Pharmacologic and Nonpharmacologic Interventions on Insomnia Symptoms and Self-reported Sleep Quality in Women With Hot Flashes: A Pooled Analysis of Individual Participant Data From Four MsFLASH Trials. Sleep. 2018 Jan 1;41(1):zsx190. doi: 10.1093/sleep/zsx190. PMID 29165623
- [Derived] Guthrie KA, LaCroix AZ, Ensrud KE, Joffe H, Newton KM, Reed SD, Caan B, Carpenter JS, Cohen LS, Freeman EW, Larson JC, Manson JE, Rexrode K, Skaar TC, Sternfeld B, Anderson GL. Pooled Analysis of Six Pharmacologic and Nonpharmacologic Interventions for Vasomotor Symptoms. Obstet Gynecol. 2015 Aug;126(2):413-422. doi: 10.1097/AOG.0000000000000927. PMID 26241433
- [Derived] Caan B, LaCroix AZ, Joffe H, Guthrie KA, Larson JC, Carpenter JS, Cohen LS, Freeman EW, Manson JE, Newton K, Reed S, Rexrode K, Shifren J, Sternfeld B, Ensrud K. Effects of estrogen and venlafaxine on menopause-related quality of life in healthy postmenopausal women with hot flashes: a placebo-controlled randomized trial. Menopause. 2015 Jun;22(6):607-15. doi: 10.1097/GME.0000000000000364. PMID 25405571
- [Derived] Ensrud KE, Guthrie KA, Hohensee C, Caan B, Carpenter JS, Freeman EW, LaCroix AZ, Landis CA, Manson J, Newton KM, Otte J, Reed SD, Shifren JL, Sternfeld B, Woods NF, Joffe H. Effects of estradiol and venlafaxine on insomnia symptoms and sleep quality in women with hot flashes. Sleep. 2015 Jan 1;38(1):97-108. doi: 10.5665/sleep.4332. PMID 25325454
- [Derived] Reed SD, Mitchell CM, Joffe H, Cohen L, Shifren JL, Newton KM, Freeman EW, Larson JC, Manson JE, LaCroix AZ, Guthrie KA. Sexual function in women on estradiol or venlafaxine for hot flushes: a randomized controlled trial. Obstet Gynecol. 2014 Aug;124(2 Pt 1):233-241. doi: 10.1097/AOG.0000000000000386. PMID 25004335
- [Derived] Joffe H, Guthrie KA, LaCroix AZ, Reed SD, Ensrud KE, Manson JE, Newton KM, Freeman EW, Anderson GL, Larson JC, Hunt J, Shifren J, Rexrode KM, Caan B, Sternfeld B, Carpenter JS, Cohen L. Low-dose estradiol and the serotonin-norepinephrine reuptake inhibitor venlafaxine for vasomotor symptoms: a randomized clinical trial. JAMA Intern Med. 2014 Jul;174(7):1058-66. doi: 10.1001/jamainternmed.2014.1891. PMID 24861828
- [Derived] Newton KM, Carpenter JS, Guthrie KA, Anderson GL, Caan B, Cohen LS, Ensrud KE, Freeman EW, Joffe H, Sternfeld B, Reed SD, Sherman S, Sammel MD, Kroenke K, Larson JC, Lacroix AZ. Methods for the design of vasomotor symptom trials: the menopausal strategies: finding lasting answers to symptoms and health network. Menopause. 2014 Jan;21(1):45-58. doi: 10.1097/GME.0b013e31829337a4. PMID 23760428

RESULTS

PARTICIPANT FLOW:
Groups:
- Low-dose 17-ß-Estradiol With Progesterone Taper: Low-dose 17-ß-estradiol oral (by mouth), 0.5 mg once per day for 8 (eight) weeks. 17-ß-estradiol is approved by the US Food and Drug Administration (FDA) and is indicated for the treatment of menopausal symptoms. ß is the Greek symbol for beta; the symbol and the word are used interchangeably. The 8 week estradiol treatment is followed 14 days (2 weeks) of progesterone taper (as medroxy-progesterone 10 mg/day).
Period: Overall Study
Arm/Group | Low-dose 17-ß-Estradiol With Progesterone Taper | Venlafaxine XR | Placebo
Started | 97 | 96 | 146
Completed | 95 | 93 | 142
Not Completed | 2 | 3 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Did not provide hot flash diary data | 1 | 3 | 3

BASELINE CHARACTERISTICS:
Population: Randomized participants per trial arm
Groups:
- Low-dose 17-ß-estradiol With Progesterone Taper: Low-dose 17-ß-estradiol: Low-dose 17-ß-estradiol oral (by mouth), 0.5 mg once per day for 8 (eight) weeks. After the 8-week treatment, women with a uterus will receive medroxyprogesterone 10 mg once per day for 2 weeks (14 days). 17-ß-estradiol is approved by the US Food and Drug Administration (FDA) and is indicated for the treatment of menopausal symptoms. ß is the Greek symbol for beta; the symbol and the word are used interchangeably.
- Total: Total of all reporting groups
Arm/Group | Low-dose 17-ß-estradiol With Progesterone Taper | Venlafaxine XR | Placebo | Total
Number analyzed (Participants) | 97 | 96 | 146 | 339
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (4.1) | 54.8 (3.7) | 54.3 (3.8) | 54.6 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 96 | 146 | 339
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 97 | 96 | 146 | 339
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.5 (6.5) | 29.3 (6.9) | 27.6 (6.8) | 28.3 (6.8)
Smoking [Number; unit: participants]
  Never | 50 | 54 | 70 | 174
  Past | 30 | 27 | 50 | 107
  Current | 17 | 14 | 24 | 55
  Missing | 0 | 1 | 2 | 3
Alcohol use (drinks/week) [Number; unit: participants]
  <7 | 71 | 77 | 117 | 265
  >=7 | 21 | 13 | 27 | 61
  Missing | 5 | 6 | 2 | 13
Marital status [Number; unit: participants]
  Never married / Divorced / Widowed | 38 | 40 | 49 | 127
  Married / living with partner | 58 | 56 | 96 | 210
  Missing | 1 | 0 | 1 | 2
Education [Number; unit: participants]
  <College graduate | 48 | 48 | 70 | 166
  College graduate | 49 | 48 | 75 | 172
  Missing | 0 | 0 | 1 | 1
Menopause status [Number; unit: participants]
  Perimenopausal | 14 | 16 | 22 | 52
  Postmenopausal | 74 | 72 | 110 | 256
  Indeterminate | 9 | 8 | 14 | 31
Years since final menstrual period (postmenopausal only) [Number; unit: participants]
  0 - 5 | 35 | 39 | 68 | 142
  6 - 10 | 23 | 20 | 29 | 72
  > 10 | 16 | 13 | 13 | 42
  Not postmenopausal | 23 | 24 | 36 | 83
Vasomotor symptom (VMS) number of participants with number of hot flashes / day [Number; unit: participants]
  < 6 | 36 | 36 | 67 | 139
  6 - < 9 | 32 | 31 | 39 | 102
  9 - < 12 | 11 | 15 | 19 | 45
  >= 12 | 18 | 14 | 21 | 53
Age at starting vasomotor symptoms (VMS), years of age [Number; unit: participants]
  < 50 | 47 | 51 | 73 | 171
  >= 50 | 48 | 44 | 71 | 163
  Missing | 2 | 1 | 2 | 5
Insomnia Severity Index (ISI) Score [Mean (Standard Deviation); unit: units on a scale] — The Insomnia Severity Index (ISI) assesses level of insomnia, an inability to sleep. There are 7 questions, each ranging in a numerical rating from 0 (zero) to 4 with 0 indicating less insomnia and 4 indicating more insomnia. The numbers from each question are summed for a total score ranging from 0 to 28 with 0 indicating less insomnia and 28 indicating more insomnia.
  units on a scale | 11.0 (6.3) | 11.7 (6.0) | 10.4 (5.8) | 11.0 (6.0)
Insomnia Severity Index (ISI) Score [Number; unit: participants]
  No clinically significant insomnia (<= 7) | 28 | 26 | 52 | 106
  Subthreshold insomnia (8 - 14) | 40 | 39 | 54 | 133
  Clinical insomnia (moderate, 15 - 21) | 21 | 25 | 32 | 78
  Clinical insomnia (severe, >= 22) | 5 | 5 | 4 | 14
  Missing | 3 | 1 | 4 | 8
Pittsburgh Sleep Quality Index (PSQI) Score [Mean (Standard Deviation); unit: units on a scale] — The Pittsburgh Sleep Quality Index (PSQI) assesses quality of sleep. There are 7 questions. Each question is scored 0 (better quality sleep) to 3 (worse quality sleep). The scores from each question are summed to a total score, ranging from 0 (better quality sleep) to 21 (worse quality sleep).
  units on a scale | 7.6 (3.6) | 7.6 (3.2) | 7.3 (3.5) | 7.5 (3.4)
Pittsburgh Sleep Quality Index (PSQI) Score [Number; unit: participants]
  Good quality sleep (< 5) | 23 | 14 | 30 | 67
  Moderate sleep quality (5 - < 8) | 21 | 35 | 46 | 102
  Poor sleep quality (>= 8) | 46 | 40 | 65 | 151
  Missing | 7 | 7 | 5 | 19
Patient Health Questionnaire (PHQ-9) Depression Score [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire (PHQ-9) assesses severity of depression. There are 10 questions with the first nine questions each scored from 0 to 3. The individual scores are summed to create a total score ranging from 0 to 45. Scores from 5 to >20 provisionally indicate, from lower to higher numbers, minimal symptoms to severe depression.
  units on a scale | 3.9 (4.4) | 3.0 (2.9) | 3.4 (3.7) | 3.4 (3.7)
PHQ-9 Depression Score [Number; unit: participants]
  No depression (0 - 4) | 68 | 70 | 108 | 246
  Mild depression (5 - 9) | 18 | 23 | 23 | 64
  Moderate depression (>= 10) | 11 | 3 | 15 | 29
Generalized Anxiety Disorder 7 (GAD-7) Score [Mean (Standard Deviation); unit: units on a scale] — Generalized Anxiety Disorder 7 (GAD-7) assesses generalized anxiety. There are 7 questions with each scored from 0 to 3. The scores from each question are summed to a total score ranging from 0 to 21. Lower scores are better.
  units on a scale | 3.0 (4.3) | 2.2 (3.0) | 2.4 (3.4) | 2.5 (3.6)
Generalized Anxiety Disorder 7 (GAD-7) Score [Number; unit: participants]
  No anxiety (0 - 4) | 73 | 76 | 116 | 265
  Mild anxiety (5 - 9) | 15 | 17 | 19 | 51
  Moderate anxiety (>= 10) | 9 | 3 | 11 | 23
Vasomotor Symptoms (VMS) as number of hot flashes [Mean (Standard Deviation); unit: Number of hot flashes per day] — Vasomotor Symptoms (VMS) frequency measures the number of hot flashes during the day and during the night. The day and night frequencies are summed for a 24-hour score.
  Number of hot flashes per day | 8.5 (5.7) | 8.2 (5.5) | 7.7 (4.8) | 8.1 (5.3)
Severity of Hot Flashes [Mean (Standard Deviation); unit: units on a scale] — Severity of hot flashes is measured as a scale from 0 to 3. Lower numbers indicate less severity and higher numbers indicate more severity.
  units on a scale | 1.1 (0.5) | 1.0 (0.5) | 1.0 (0.4) | 1.0 (0.5)
Bothersomeness of Hot Flashes [Mean (Standard Deviation); unit: units on a scale] — Bothersomeness of hot flashes is measured on a scale from 0 to 3. Lower numbers indicate less bother and higher numbers indicate more bother.
  units on a scale | 2.1 (0.5) | 2.0 (0.5) | 2.0 (0.5) | 2.0 (0.5)
Perceived Hot Flash Interference (Hot Flash Related Daily Interference Scale; HFRDIS) [Mean (Standard Deviation); unit: units on a scale] — The perceived hot flash related daily interference scale (HFRDIS) is a tool for assessing the impact of hot flashes on quality of life. There are 10 questions with each having a score ranging from 0 to 10. The scores from each question are summed for a total score ranging from 0 to 100. Lower numbers indicate less interference and higher numbers indicate more interference.
  units on a scale | 36.9 (23.8) | 36.8 (23.4) | 32.8 (21.3) | 35.1 (22.6)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Hot Flashes (Vasomotor Symptom [VMS] Frequency) -- Week 4
Description: Measured by self-report diary twice daily (day and night). The day and night frequencies were summed to produce a single number of hot flashes per day. The single number of hot flashes per day were summed and averaged for one week prior to the week 4 study assessment to produce a mean daily frequency for week 4.
Time Frame: Week 4
Population: Intention-to-treat, i.e., all participants with follow-up data were included.
Measure: Mean (95% Confidence Interval); unit: number of hot flashes per day
Arm/Group | Low-dose 17-ß-estradiol With Progesterone Taper | Venlafaxine XR | Placebo
Number analyzed (Participants) | 91 | 93 | 139
number of hot flashes per day | 5.3 [4.2 to 6.5] | 5.1 [4.1 to 6.0] | 5.8 [4.9 to 6.7]

2. Secondary Outcome: Severity of Hot Flashes -- Week 4
Description: Measured by self-report diary twice daily (day and night) for 7 days. Severity ratings ranged from 0 to 3 with lower numbers being less severe and higher numbers being more severe. Data from the day and night severity ratings were averaged for a single daily score. The single daily scores for the week prior to the week 4 study assessment were summed and averaged to produce a mean daily VMS severity for week 4.
Time Frame: Week 4
Population: Intention-to-treat, i.e., all participants with follow-up data were included.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Low-dose 17-ß-estradiol With Progesterone Taper | Venlafaxine XR | Placebo
Number analyzed (Participants) | 81 | 86 | 134
units on a scale | 0.7 [0.6 to 0.9] | 0.7 [0.5 to 0.8] | 0.8 [0.7 to 0.9]

3. Secondary Outcome: Severity of Hot Flashes -- Week 8
Description: Measured by self-report diary twice daily (day and night) for 7 days. Severity ratings ranged from 0 to 3 with lower numbers being less severe and higher numbers being more severe. Data from the day and night severity ratings were averaged for a single daily score. The single daily scores for the week prior to the week 8 study assessment were summed and averaged to produce a mean daily VMS severity for week 8.
Time Frame: Week 8
Population: Intention-to-treat, i.e., all participants with follow-up data were included.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Low-dose 17-ß-estradiol With Progesterone Taper | Venlafaxine XR | Placebo
Number analyzed (Participants) | 73 | 86 | 133
units on a scale | 0.6 [0.4 to 0.7] | 0.6 [0.4 to 0.7] | 0.7 [0.6 to 0.8]
Statistical Analysis 1: Comparison: Low-dose 17-ß-estradiol With Progesterone Taper vs Placebo; Outcome differences between active treatment and placebo; Test type: Superiority or Other; p = 0.02, repeated measures linear model — P-values from active treatment vs. placebo contrasts in a repeated measures linear model of outcome as a function of treatment arm, clinical site, week, and baseline outcome. The a priori threshold for statistical significance was 0.025; Robust standard errors were calculated using generalized estimating equations to account for within-participant correlation between repeated measures
Statistical Analysis 2: Comparison: Venlafaxine XR vs Placebo; Outcome differences between active treatment and placebo; Test type: Superiority or Other; p = 0.02, repeated measures linear model — p-values from active treatment vs. placebo contrasts in a repeated measures linear model of outcome as a function of treatment arm, clinical site, week, and baseline outcome. The a priori threshold of statistical significance was 0.025; [statistical method as in outcome 3, analysis 1]

4. Primary Outcome: Frequency of Hot Flashes (Daily Vasomotor Symptom [VMS] Frequency) -- Week 8
Description: Measured by self-report diary twice daily (day and night). The day and night frequencies were summed to produce a single number of hot flashes per day. The single number of hot flashes per day were summed and averaged for one week prior to the week 8 study assessment to produce a mean daily frequency for week 8.
Time Frame: Week 8
Population: Intention-to-treat, i.e., all participants with follow-up data were included.
Measure: Mean (95% Confidence Interval); unit: number of hot flashes per day
Arm/Group | Low-dose 17-ß-estradiol With Progesterone Taper | Venlafaxine XR | Placebo
Number analyzed (Participants) | 92 | 89 | 137
number of hot flashes per day | 3.9 [2.9 to 4.9] | 4.4 [3.5 to 5.3] | 5.5 [4.7 to 6.3]
Statistical Analysis 1: Comparison: Low-dose 17-ß-estradiol With Progesterone Taper vs Placebo; VMS frequency values were log transformed for modeling; Test type: Superiority or Other; p < 0.001, repeated measures linear model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Venlafaxine XR vs Placebo; VMS frequency values were log transformed for modeling; Test type: Superiority or Other; p = 0.005, repeated measures linear model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]

5. Secondary Outcome: Bothersomeness of Hot Flashes -- Week 4
Description: Measured by self-report diary twice daily (day and night) for 7 days. Bothersomeness ratings ranged from 0 to 3 with lower numbers being less bothersome and higher numbers being more bothersome. Data from the day and night bothersomeness ratings were averaged for a single daily score. The single daily scores for the week prior to the week 4 study assessment were summed and averaged to produce a mean daily VMS bothersomeness for week 4.
Time Frame: Week 4
Population: Intention-to-treat, i.e., all participants with follow-up data were included.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Low-dose 17-ß-estradiol With Progesterone Taper | Venlafaxine XR | Placebo
Number analyzed (Participants) | 82 | 88 | 135
units on a scale | 1.6 [1.4 to 1.7] | 1.6 [1.4 to 1.7] | 1.7 [1.6 to 1.8]

6. Secondary Outcome: Bothersomeness of Hot Flashes -- Week 8
Description: Measured by self-report diary twice daily (day and night) for 7 days. Bothersomeness ratings ranged from 0 to 3 with lower numbers being less bothersome and higher numbers being more bothersome. Data from the day and night bothersomeness ratings were averaged for a single daily score. The single daily scores for the week prior to the week 8 study assessment were summed and averaged to produce a mean daily VMS bothersomeness for week 8.
Time Frame: Week 8
Population: Intention-to-treat, i.e., all participants with follow-up data were included.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Low-dose 17-ß-estradiol With Progesterone Taper | Venlafaxine XR | Placebo
Number analyzed (Participants) | 73 | 86 | 133
units on a scale | 1.4 [1.2 to 1.6] | 1.4 [1.3 to 1.6] | 1.6 [1.5 to 1.7]
Statistical Analysis 1: Comparison: Low-dose 17-ß-estradiol With Progesterone Taper vs Placebo; Outcome differences between active treatment and placebo; Test type: Superiority or Other; p = 0.01, repeated measures linear model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Venlafaxine XR vs Placebo; Outcome differences between active treatment and placebo; Test type: Superiority or Other; p = 0.07, repeated measures linear model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]

7. Secondary Outcome: Perceived Hot Flash Interference (Hot Flash Related Daily Interference Scale; HFRDIS) -- Week 4
Description: The perceived hot flash related daily interference scale (HFRDIS) is a tool for assessing the impact of hot flashes on quality of life. There are 10 questions with each having a score ranging from 0 to 10. The scores from each question are summed for a total score ranging from 0 to 100. Lower numbers indicate less interference and higher numbers indicate more interference.
Time Frame: Week 4
Population: Intention-to-treat, i.e., all participants with follow-up data were included.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Low-dose 17-ß-estradiol With Progesterone Taper | Venlafaxine XR | Placebo
Number analyzed (Participants) | 84 | 83 | 128
units on a scale | 18.3 [13.8 to 22.8] | 19.8 [15.6 to 23.9] | 24.2 [20.7 to 27.7]

8. Secondary Outcome: Perceived Hot Flash Interference (Hot Flash Related Daily Interference Scale; HFRDIS) -- Week 8
Description: as for outcome 7
Time Frame: Week 8
Population: Intention-to-treat, i.e., all participants with follow-up data were included.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Low-dose 17-ß-estradiol With Progesterone Taper | Venlafaxine XR | Placebo
Number analyzed (Participants) | 92 | 86 | 137
units on a scale | 14.6 [10.6 to 18.7] | 18.3 [13.8 to 22.7] | 21.5 [18.1 to 24.9]
Statistical Analysis 1: Comparison: Low-dose 17-ß-estradiol With Progesterone Taper vs Placebo; Outcome differences between active treatment and placebo; Test type: Superiority or Other; p < 0.001, repeated measures linear model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Venlafaxine XR vs Placebo; Outcome differences between active treatment and placebo; Test type: Superiority or Other; p = 0.03, repeated measures linear model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: At 1-, 4, and 8-weeks, potential adverse events were assessed by a Management and Safety Interview. Symptoms data were collected at screening and weeks 4 and 8. Data are reported as newly emergent adverse events.
Groups:
- Low-dose 17-ß-estradiol: Low-dose 17-ß-estradiol: Low-dose 17-ß-estradiol oral (by mouth), 0.5 mg once per day for 8 (eight) weeks. After the 8-week treatment, women with a uterus will receive medroxyprogesterone 10 mg once per day for 2 weeks (14 days). 17-ß-estradiol is approved by the US Food and Drug Administration (FDA) and is indicated for the treatment of menopausal symptoms. ß is the Greek symbol for beta; the symbol and the word are used interchangeably.
Arm/Group | Low-dose 17-ß-estradiol | Venlafaxine XR | Placebo
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/96 | 0/146
Other Adverse Events (participants affected / at risk) | 53/97 | 65/96 | 88/146
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Low-dose 17-ß-estradiol (N=97) | Venlafaxine XR (N=96) | Placebo (N=146)
Any fatigue/arousal symptom (General disorders) | 20/85 | 26/81 | 33/127
Any central nervous system symptom (Nervous system disorders) | 22/92 | 30/94 | 36/142
Any GI symptom (Gastrointestinal disorders) | 23/94 | 25/93 | 44/142
Breast tenderness (Reproductive system and breast disorders) | 5/90 | 0/93 | 8/142
Vaginal secretions (Reproductive system and breast disorders) | 2/90 | 3/90 | 3/139
Any musculoskeletal symptom (Musculoskeletal and connective tissue disorders) | 9/92 | 5/94 | 13/141
Any miscellaneous symptom (General disorders) | 28/94 | 36/94 | 43/142

LIMITATIONS AND CAVEATS:
Findings may be specific to the particular dose of each agent used, treatment period, as well as the preparation and oral administration of estrogen therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No